CLINICAL TRIAL: NCT03156907
Title: High Dosage Buprenorphine as a Drug Strategy Withdrawal Assistance of Analgesics Opioid After Failure of an Opioid Tapering-off Strategy.
Brief Title: High Dosage Buprenorphine as a Drug Strategy Withdrawal Assistance of Analgesics Opioid
Acronym: SEVROP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-325; 2015-003173-15 (Other: 2015-003173-15)
Record Dates: First submitted 2017-05-05; First posted 2017-05-17 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: High Dosage Buprenorphine
Keywords: High dosage Buprenorphine (HDB); Chronic pain; Analgesics opioids; Withdrawal symptoms
MeSH Terms: conditions — Chronic Pain; Substance Withdrawal Syndrome | interventions — Buprenorphine

STUDY DESIGN:
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic pain patients (Experimental): The primary objective of this study is to assess the success rate at 6 months of opioid temporary rotation by High Dosage Buprenorphine (HDB) taper dose in chronic non cancer pain patients (CNCP) with physical withdrawal symptoms making opioid withdrawal impossible.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — HDB is started (J0) at the dosage of 4 mg/ day (with a possible adjustment ± 2 mg at 24h, depending on the patient withdrawal symptoms intensity or tolerance).

SUMMARY:
The prevalence of analgesics opioids addiction in chronic pain patient is very difficult to know. Many studies indicated that the prevalence of addiction varied from 0% up to 50% in chronic non cancer pain patients, and from 0% up to 7.7% in cancer pain patients. Analgesics opioids use have increasingly been increased in chronic pain for 20 years. However, a long use, at least 3 months in this type of pain has not proved a large efficiency and we have noticed a habituation, tolerance and withdrawal when treatment was decreased or stopped. In current practice, patients with chronic pain, often keep their analgesics opioids despite the absence of pain relief and benefits in quality of life.

Nowadays, no withdrawal strategy is the reference in chronic non-cancer pain patients with physical opioid dependence. The most common clinical strategy is progressive decrease of analgesic opioid. But this strategy is often a failure in these patients (no data are available in literature).

It's necessary to make a prospective pilot study to assess benefits from this practice.

The primary objective of this study is to assess a new ambulatory withdrawal strategy, consisting of a temporary opioid rotation with buprenorphine in CNCP patients suffering from physical withdrawal symptoms and who have failed a conventional strategy of progressive withdrawal from their opioid analgesic treatment.

DETAILED DESCRIPTION:
This study is designed as a type 2 multicenter clinical trial combining 3 Pain Clinics.

Patients were consecutively recruited from the active file of 3 Pain Clinics in France (Clermont-Ferrand, Vichy and le Puy-en-Velay). Patients meeting all inclusion criteria were enrolled after receiving oral and written information about the study and after obtaining written informed consent.

At baseline, they completed 5 questionnaires including: Brief Pain Inventory (BPI), Hospital Anxiety and Depression scale (HAD), Leeds sleep Evaluation Questionnaire (LSEQ), Short version of Short Form 36 Health Survey (SF 12), Clinical Opioid Withdrawal Scale (COWS) and underwent 2 tests with algometer and pupillometer. After inclusion, all patients started an opioid tapering-off protocol (Figure 1, Step 1) according to a standardized scheme of opioid gradual decrease defined by 3 medical experts in addictology, pain management and pharmacology.

Step 1 (from inclusion to 3 months): Patients will start to taper off their opioid dose according to a specific schedule. They will be seen by a physician on a monthly basis and contacted by phone 48-72h after each decrease in opioid dosage to detect withdrawal symptoms using the COWS specific scale. After 3 months, all patients who fail the opioid tapering-off protocol will be included in a non-responder group, while the others who succeed the withdrawal protocol will be included in a responder group:

* A responder will be defined by strict adherence to the schedule leading to a 50% reduction in the initial daily dose of opioid after 3 months. In this case, patients will continue with step 1 and decrease their opioid dose according to the same withdrawal protocol. They will be seen by a physician on a monthly basis and contacted by phone 48-72h after each stage of opioid dose reduction, until the opioid treatment is completely discontinued after 6 months of the withdrawal protocol. At 6 months, patients will fill out the same questionnaires and perform the same tests as at the baseline visit. Finally, after 9 months, patients will be contacted by phone to check that withdrawal is being maintained and to collect data on ongoing analgesic treatment.
* A non-responder will be defined as a failure of the withdrawal protocol, by non-compliance with the schedule, leading to a 50% reduction in the initial daily dose of opioid treatment after 3 months or when tapering off fails, leading the patient to re-increase the opioid dose. Thus, these patients will proceed to step 2 and start temporary rotation with buprenorphine.

Step 2:

* From D0 to D0+28 days - buprenorphine treatment/stabilization Buprenorphine will be administered initially (D0) for 28 days at a dose of 4 mg/day (possible adjustment of ±2mg/day with the possibility to increase the dose up to 8 mg/day during the first 24-48 hours, depending on the severity of withdrawal symptoms or patient tolerance). Questionnaires (BPI, HADS, LSEQ, SF-12, COWS) and tests (algometer and pupillometer) will be completed at D0, and the physician will assess the efficacy and safety of buprenorphine by phone call at D0 + 24h/48 h and at D0 + 7 days.
* From D0 + 28 days to D0 + 9th month after rotation by buprenorphine The buprenorphine treatment will be tapered off in 1 mg steps every 28 days until the complete cessation of buprenorphine after 9 months of withdrawal. Patients will be seen by a physician every 28 days and will be contacted by phone 48-72h after each decrease in the buprenorphine dose. The COWS questionnaires and a pain assessment (11-point NRS) will be completed at each medical consultation.
* D0 + 9th month A urine opioid test (primary outcome) will be performed to validate the total opioid withdrawal (including buprenorphine). Patients will complete different questionnaires (BPI, HADS, LSEQ, SF 12, COWS) and perform different tests (algometer and pupillometer).
* Follow-up phone call at 12 months The patients will be contacted by phone to check on their continued withdrawal and ongoing analgesic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years,
* patients with CNCP who have been treated for more than 6 months with a single opioid analgesic (weak or strong; long acting and/or immediate release),
* Patients will be required to have an indication to stop or reduce opioid therapy (i.e. unfounded indication, tolerance, ineffectiveness, and/or adverse effects), and/or have physical withdrawal symptoms between opioid administrations (Clinical Opioid Withdrawal Scale (COWS) assessment),
* Patients must have given their comprehensive informed consent and be affiliated with the French social security system.

Exclusion Criteria:

* not have an opioid use disorder with craving (assessment by investigator according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)) or misuse (assessment by the Prescription Opioid Misuse Index (POMI)[28]) related to opioid use,
* ongoing treatment with ketamine,
* chronic cancer pain,
* contraindication to buprenorphine (hypersensitivity to an active substance or its excipients, severe hepatic and/or respiratory dysfunction, alcohol use disorder or delirium tremens),
* alcohol use disorder,
* pregnant or breastfeeding,
* involved in any other interventional trial, or be subject to legal protection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Absence of opioid in urine test after rotation by HDB | Month 6
  Validating total opioid withdrawal (including HDB)

SECONDARY OUTCOMES:
Rate of opioid tapering-off protocol success by decrease of 50% of initial posology | Month 3
Rate of opioid tapering-off protocol success by total taper opioid withdrawal | Month 6
The pain will be assessed by the questionnaire Brief pain Inventory (BPI) | Day 1, Month 1, Month 6
The quality of life will be assessed by questionnaire SF12 (Short version of Short Form 36 Health Survey) | Day 1, Month 1, Month 6
The anxiety and depression will be assessed by questionnaire HAD (Hospital anxiety and depression scale) | Day 1, Month 1, Month 6
The sleep will be assessed by questionnaire LSEQ (Leeds sleep evaluation questionnaire) | Day 1, Month 1, Month 6
Evaluation of the correlation between pupillary dilation (pupillometer) and pain (NRS 0-10). | Day 1, Month 1, Month 6
Evaluation of pain intensity (NRS 0-10) by the pressure algometry measurement. | Day 1, Month 1, Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Bertin C, Kerckhove N, Ferrer F, Pereira B, Duale C, Richard D, Authier N, Delage N. Buprenorphine Substitution as a Tapering Strategy for Opioid Discontinuation in Patients with Chronic Pain: A Nonrandomized and Proof of Concept Study. Pain Ther. 2025 Dec;14(6):1783-1795. doi: 10.1007/s40122-025-00781-z. Epub 2025 Oct 3. PMID 41042438